CLINICAL TRIAL: NCT03627052
Title: A Phase 2, Double-Blind, Dose-Ranging, Placebo-Controlled Study With Open-Label Extension to Evaluate the Safety and Efficacy of Itacitinib in Moderate to Severe Ulcerative Colitis
Brief Title: A Study to Evaluate the Safety and Efficacy of Itacitinib in Moderate to Severe Ulcerative Colitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn due to lack of recruitment. No patients enrolled. No safety concerns.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 39110-210
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Moderate to Severe Ulcerative Colitis
Keywords: Inflammatory bowel disease; ulcerative colitis; Janus kinase inhibitor; JAK1
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — itacitinib; INCB039110

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Itacitinib (Experimental)
  Interventions: Drug: Itacitinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itacitinib — In the double-blind period, itacitinib administered orally once or twice daily at the protocol-defined dose according to treatment group randomization. In the open-label extension, itacitinib administered at doses determined from the double-blind period.
  Other Names: INCB039110
  Arms: Itacitinib
Drug: Placebo — Placebo administered orally twice daily in the double-blind period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of itacitinib in participants with moderate to severe ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of UC at least 12 weeks before screening based on clinical, endoscopic, and histopathological evidence.
* Have a 3-component Mayo score of 4 to 9, which includes a modified Mayo Endoscopy Score (mMES) of ≥ 2 as determined by a central reader, a rectal bleeding score of ≥ 1, and a stool frequency score of ≥ 1.
* Must have failed or be intolerant to (discontinued the medication due to an adverse event as determined by the investigator) at least 1 of the following treatments for UC: Oral corticosteroids, azathioprine or 6-mercaptopurine, biologic therapy (eg, infliximab, vedolizumab or adalimumab).
* Participants currently receiving the following treatment(s) for UC are eligible, provided they have been receiving acceptable and stable dose(s): oral 5-ASA or oral corticosteroids.
* No evidence of active or latent or inadequately treated tuberculosis infection.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Clinical signs of fulminant colitis or toxic megacolon.
* Presence of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, or clinical or radiographic findings suggestive of Crohn's disease.
* Disease limited to the distal 15 cm of the colon.
* Receiving (or expected to receive) the following therapies within protocol-designated timeframes before the baseline visit or during the study: Natalizumab; anti-TNF therapy; Vedolizumab or any investigational anti-adhesion molecule therapy; Ustekinumab or any on or off label biologic therapy; interferon therapy; cyclosporine, mycophenolate, or tacrolimus; daily dose of oral corticosteroids ≥ 25 mg prednisone or equivalent; intravenous corticosteroids; rectally administered formulation of corticosteroids or 5-aminosalicylic acid; and AZA, 6-MP, or methotrexate.
* Enema treatments within 2 weeks of the baseline visit, with the exception of enema bowel preparations for clinical assessments.
* Positive stool examinations for enteric pathogens, pathogenic ova or parasites, or Clostridium difficile toxin at the screening visit.
* Other immunocompromised states and history of opportunistic infections.
* History of stomach or intestinal surgery, including bariatric surgery (Note: appendectomy and/or cholecystectomy, is allowed).

  o surgery for UC or likely to require surgery for UC during the study.
* If at risk for colorectal cancer, must have had a colonoscopy within protocol-defined timeframes.
* History of recurrent, disseminated, or multiple dermatomal herpes zoster.
* History of alcohol or drug abuse.
* History of active malignancy within 5 years of screening, excluding superficial basal and squamous cell carcinoma of the skin and adequately treated carcinoma in situ of the cervix.
* Current or recent history (within 30 days before randomization) of a clinically meaningful viral, bacterial, fungal, parasitic, or mycobacterial infection.
* Previously received either lymphocyte apheresis or selective monocyte granulocyte apheresis (eg, Cellsorba) within 1 year of baseline.
* History of unstable ischemic heart disease or uncontrolled hypertension.
* Positive serology test results for HIV, for hepatitis B surface antigen or core antibody, or for HCV antibody with detectable RNA at screening.
* Participants taking potent systemic CYP3A4 inhibitors or inducers or fluconazole within 2 weeks or 5 half-lives (whichever is longer) of baseline.
* Participants taking P-gp substrates with narrow therapeutic index, including digoxin within 2 weeks or 5 half-lives (whichever is longer) of baseline.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a Clinical Response | Week 8
  To evaluate the efficacy of itacitinib inducing a Clinical Response.

SECONDARY OUTCOMES:
Proportion of participants with Endoscopic Response | Week 8
  To evaluate the efficacy of itacitinib on endoscopic outcomes.
Proportion of participants with Mucosal Healing | Week 8
  To evaluate the efficacy of itacitinib on endoscopic outcomes.
Proportion of participants in Endoscopic Remission | Week 8
  To evaluate the efficacy of itacitinib on endoscopic outcomes.
Proportion of participants in Clinical Remission | Week 8
  To evaluate the efficacy of itacitinib on clinical outcomes.
Change from baseline in 3-component Mayo score | Week 8
  To evaluate the efficacy of itacitinib on clinical outcomes.
Change from baseline in Physician's Global Assessment score | Week 8
  To evaluate the efficacy of itacitinib on clinical outcomes.
Change in Quality of Life score as measured by the Inflammatory Bowel Disease Questionnaire (IBDQ) | Week 8
  To evaluate the efficacy of itacitinib on quality of life outcomes.
Cmax of itacitinib | Week 4
  Maximum observed plasma concentrations.
Ctau of itacitinib | Weeks 2 and 4
  Plasma concentrations
Stool concentration of itacitinib -~30-hr collection | Week 4
Number of treatment-emergent adverse events | Up to approximately 60 weeks
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Brown, MD, Study Director — Incyte Corporation

IPD SHARING:
Plan to Share IPD: No